CLINICAL TRIAL: NCT03641612
Title: Effect of Different Root Canal Instruments on Removal of Endotoxins From Necrotic Root Canals (A Randomized Clinical Trial)
Brief Title: Effect of Different Root Canal Instruments on Removal of Endotoxins From Necrotic Root Canals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heba Elasfouri (Other)
Responsible Party: Sponsor-Investigator, Heba Elasfouri, lecturer of endodontics- faculty of dentistry- cairo university, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CEBD-CU-2018-8-17
Record Dates: First submitted 2018-08-16; First posted 2018-08-22 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Endodontic Disease
Keywords: rotary instruments; endotoxins
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Intervention Model Description: The trial design of this study will be a prospective, parallel, Randomized clinical trial (RCT).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one shape (Experimental): single file rotary system
  Interventions: Other: one shape
- protaper next (Active Comparator): multiple file rotary system
  Interventions: Other: protaper next

INTERVENTIONS:
Other: one shape — canal fluid sample before and after root canal instrumentation
  Arms: one shape
Other: protaper next — canal fluid sample before and after root canal instrumentation
  Arms: protaper next

SUMMARY:
• Grouping: The patients will be randomly assigned into two equal groups Group : OneShape Group: ProtaperNext

* Endodontics procedure steps:

  1. Patient will be anesthetized by using infiltration local anesthesia or nerve block according to the tooth location in mandibular or maxillary arch respectively.
  2. All caries will be removed, then isolation using rubber dam, the crown and surrounding structures will be disinfected with 30% H2O2( hydrogen peroxide) for 30 seconds, followed by 2.5% NaOCl for the same period of time and then inactivated with 5% sodium thiosulphate.

  2- For the access cavity preparation, a sterile/apyrogenic high-speed diamond bur will be used in conjunction with manual irrigation with sterile saline. Before entering the pulp chamber, the access cavity will be disinfected according to the protocol described above.

  2- Root canal length will be determined, by preoperative radiograph then (S1) will be taken by introducing a sterile/apyrogenic paper point #15/ 20 (5paper points) into the full length of the canal and left there for 1 minute. Then, the sample will be placed in an apyrogenic glass and stored in -20°. Then canal length will be confirmed by apex locator.

  3- Cleaning and shaping will be done using either One shape or Protaper next rotary instruments in crown down preparation technique with the use of in an endodontic motor according to the manufacturer instructions, the canals will be thoroughly irrigated using 3ml of 2.5% Sodium hypochlorite between every subsequent instrument.

  4-After root canal preparation, NaOCl will be inactivated with 5 mL of sterile 5% sodium thiosulphate for 1 minute, which then will be removed with 5 mL of sterile/apyrogenic saline solution., which then will be removed with 5 mL of sterile/apyrogenic saline solution. second endotoxin sample (S2) will be taken from the root canals. (5 paper point size of the master cone).

  5- After completion of instrumentation and irrigation, obturation will be done using size 30/ 0.4 taper gutta-percha cones and auxiliaries as needed using the modified single cone technique.

Determination of Endotoxin Concentration Human endotoxin (ET) ELISA Kit will be used to measure endotoxin concentrations in the root canals before and after chemomechanical procedures.

DETAILED DESCRIPTION:
Materials and Methods:

A. Trial Design:

The trial design of this study will be a prospective, parallel, Randomized clinical trial (RCT). The clinical trial involves research using human participants. In this trial, the participants will be randomly allocated to receive one of two interventions according to the protocol created by the investigator; one of these interventions will be the control. The investigator is to determine the safety and/or the efficacy of the interventions after being received by the participants by measuring the outcomes because the outcomes will be measured, RCTs are quantitative studies.

• Grouping: The patients will be randomly assigned into two equal groups according to the type of rotary endodontic system used during root canal preparation: Group : OneShape Group : ProtaperNext

* Endodontics procedure steps:

  1. Patient will be anesthetized by using infiltration local anesthesia or nerve block according to the tooth location in mandibular or maxillary arch respectively.
  2. All caries will be removed, then isolation using rubber dam, the crown and surrounding structures will be disinfected with 30% H2O2 ( hydrogen peroxide) for 30 seconds, followed by 2.5% NaOCl for the same period of time and then inactivated with 5% sodium thiosulphate.

  2- For the access cavity preparation, a sterile/apyrogenic high-speed diamond bur will be used in conjunction with manual irrigation with sterile saline. Before entering the pulp chamber, the access cavity will be disinfected according to the protocol described above.

  2- Root canal length will be determined, by preoperative radiograph then (S1) will be taken by introducing a sterile/apyrogenic paper point #15/ 20 (5paper points) into the full length of the canal and left there for 1 minute. Then, the sample will be placed in an apyrogenic glass and stored in -20°. Then canal length will be confirmed by apex locator.

  3- Cleaning and shaping will be done using either One shape or Protaper next rotary instruments in crown down preparation technique with the use of in an endodontic motor according to the manufacturer instructions, the canals will be thoroughly irrigated using 3ml of 2.5% Sodium hypochlorite between every subsequent instrument.

  4-After root canal preparation, NaOCl will be inactivated with 5 mL of sterile 5% sodium thiosulphate for 1 minute, which then will be removed with 5 mL of sterile/apyrogenic saline solution., which then will be removed with 5 mL of sterile/apyrogenic saline solution. second endotoxin sample (S2) will be taken from the root canals. (5 paper point size of the master cone).

  5- After completion of instrumentation and irrigation, obturation will be done using size 30/ 0.4 taper gutta-percha cones and auxiliaries as needed using the modified single cone technique.

  6- All procedures will be done in a single-visit, checked radiographically and recorded in the procedure chart.

Determination of Endotoxin Concentration Human endotoxin (ET) ELISA Kit will be used to measure endotoxin concentrations in the root canals before and after chemomechanical procedures.

As a parameter for calculation of the amount of endotoxins in the root canal samples, a standard curve will be plotted by using the endotoxin of known concentration supplied by the kit according to the manufacturer's instructions.

The test procedure will be performed according to the manufacturer's instructions. And the absorbance of endotoxins will be measured by using spectrophotometer at wavelength 450 nm.

D. Outcomes:

Evaluation of the antibacterial effect of using One Shape and Protaper Next rotary endodontic NiTi instruments for root canal preparation using Human endotoxin (ET) ELISA Kit

E. Randomization:

The randomization will be done in three steps:

1. Sequence generation:

   The random sequence generation will be done for the patients' numbers (from 1 to 38) using Microsoft Excel software.

   Allocation concealment mechanism:

   The allocation concealment will be phone-based.
2. Implementation:

The random sequence will be done by a colleague and the random sequence table will be kept with him. After eligibility assessment, the operator would call the colleague for eligibility checking and to know the group assignment for the patients.

F. Blinding:

Participants, outcome assessor and data analyst will be blinded in this trial. The operator will be not blinded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are medically free and good health.
* Patient 's age between 20-60years.
* Patients with posterior teeth diagnosed clinically and confirmed by thermal sensitivity tests as teeth with necrotic pulp.
* Positive patient's acceptance for participation in the study.

Exclusion Criteria:

* -Pregnancy or lactation
* Medically compromised patients -Patients aged less than20 or more than 60 years.-
* Patients unable to give informed consent.
* Previous endodontic therapy of the affected tooth .
* Teeth diagnosed with vital pulp.
* Teeth with periodontal pocket more than 3mm deep.
* Teeth with abnormal anatomy and calcified canals.
* Teeth with caries below the bony level (non-restorable tooth).
* Teeth with periapical swelling or sinus tract.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
endotoxin change | Samples will be collected before and after chemomechanical preparation over 2 months
  Human endotoxin (ET) ELISA Kit will be used to measure endotoxin concentrations in the root canals before and after chemomechanical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: heba elasfouri, lecturer, Principal Investigator — Cairo University; marwa bedier, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University Faculty of Dentistry, Cairo, Egypt